CLINICAL TRIAL: NCT07215897
Title: Evaluating Covered California's Grocery Support Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Covered California (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-42548; 21-C027-11 (Other Grant/Funding Number: Covered California)
Record Dates: First submitted 2025-10-07; First posted 2025-10-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Chronic Conditions, Multiple; Chronic Conditions; Food Insecurity; Low-Income Population
Keywords: chronic conditions; food insecurity; grocery benefit; low-income
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Intervention Model Description: Participants (n=6,975) were randomized into the intervention n=3,486) or active comparator (n=3,489) stratified by preferred language (English vs. non-English) and Covered California metal tier (Silver vs. Bronze). The intervention consists of a monthly or lump sum grocery support program provided in the form of a reloadable cash card usable at food retailers including those that sell non-food items.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Monthly grocery support program (Experimental): The intervention entails the provision of an $80 monthly payment (adjusted by household size) in the form of a re-loadable cash card to be used at food retailers including food retailers who sell non-food item.
  Interventions: Other: Grocery Support Monthly Program
- One-time grocery support payment (Active Comparator): At the end of the study period (12 months), active comparator participants are provided a lump sum payment of $960 (adjusted by household size) as a re-loadable cash card to use at food retailers. No intervention is provided during the 12-month evaluation period.
  Interventions: Other: Grocery Support One-Time Payment

INTERVENTIONS:
Other: Grocery Support Monthly Program — $80 monthly (adjusted by household size), re-loadable cash card for use at food retailers to purchase fresh and packaged foods, baby food and formula, and/or non-alcoholic drinks
  Arms: Monthly grocery support program
Other: Grocery Support One-Time Payment — No intervention is provided during the 12-month evaluation period. A $960 one-time (adjusted by household size) cash card for use at food retailers provided after the 12 month evaluation period to purchase fresh and packaged foods, baby food and formula, and/or non-alcoholic drinks
  Arms: One-time grocery support payment

SUMMARY:
This is a pragmatic randomized controlled trial (RCT) of Covered California's Grocery Support Program. This pragmatic RCT will test the efficacy of providing a monthly food card benefit for adults with food insecurity, a chronic condition, and incomes below 250% of the federal poverty level (FPL) compared with a group who receives a lump sum payment.

DETAILED DESCRIPTION:
In 2024, Covered California initiated multiple Population Health Investments (PopHIs) based on funds collected by participating plans if they failed to meet a set of quality benchmarks related to diabetes control, blood pressure control, colorectal cancer screening, and childhood immunizations. One priority area for the PopHIs was food insecurity among patients who manage chronic diseases. Food insecurity, defined by the United States Department of Agriculture (USDA) as a "lack of access to enough food for an active, healthy life" effects 18% of newly enrolled Covered California members. Food insecurity is more pronounced and is associated with poor clinical outcomes and more avoidable and costly healthcare utilization among individuals who manage chronic disease. The burden of disease is high among Covered California members; for every 1,000 Covered California enrollees with one or more years of continuous enrollment, 390 have a chronic disease diagnosis. The goal of the proposed research is to evaluate the impact of a 12-month grocery support program on participant food insecurity and other outcomes compared to a single payment at the end of 12 months. Participants were invited to enroll in the program if they were active members of Covered California at the time of enrollment, and had 1) a documented chronic condition, 2) food insecurity measured using the validated two-item screener), and 3) an income at or below 250% of the FPL. Participants were randomly assigned to receive either an $80 reusable semi-restricted cash card re-loaded monthly for one year or a one-time cash card of $960 (payments in both arms adjusted based on household size). Retailers are restricted to food retailers, which includes retailers that do sell non-food goods. The study has four main data sources: survey data from surveys repeated at baseline and 12-months; cash card spending data; qualitative participant interview data and claims data.

Specific Aims are to:

Aim 1 - To evaluate the impact of the grocery support program on participant food insecurity and other dietary outcomes.

H1: Participants who receive the monthly payment will have decreased rates of food insecurity and improved dietary outcomes 12-months after participating compared to participants who do not receive the monthly payment.

Aim 2 - To assess the impact of the grocery support program on self-rated health, healthcare experiences, and social risks and other quality of life measures.

H1: Participants who receive the monthly payment will have improved self-rated health, healthcare experiences, and quality of life, and fewer social risks compared to participants who do not receive the monthly payment.

Aim 3 - To analyze the impact of the grocery support program on participant's health utilization and outcomes.

H1: Relative to participants who do not receive the monthly payment, Grocery Support Program participants will have fewer hospitalizations and Emergency Department (ED) visits and more primary care visits.

H2: Relative to participants who do not receive the monthly payment, Grocery Support Program participants will have greater improvements in chronic disease clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

Members of the household are eligible to participate if the recruited participant:

* Active Covered California member
* Adult >= 18 years of age
* Has a chronic condition identifiable in Covered California's medical claims
* Screened positive for food insecurity via 2-item Hunger Vital Sign
* Income <250% federal poverty level

Exclusion Criteria:

* Negative for food insecurity via 2-item Hunger Vital Sign
* Income ≥250% federal poverty level

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6975 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in food insecurity status | Baseline, 12 months
  Measured by 2-item Hunger Vital Sign, a validated tool to assess food insecurity. Responses that indicate that food sometimes or often did not last or ran out before the end of the month indicate food insecurity

SECONDARY OUTCOMES:
Change in nutrition security | Baseline, 12 months
  Measured using the one-item response allowing calculation of the proportion of participants that report difficulty getting and eating healthy foods.
Change in diet quality | Baseline, 12 months
  Measured using the self-reported number of servings of vegetables or number of days where higher fat foods were consumed during the past 7 days, by study arm
Proportion of participants with acute health care utilization | 2 years before study start until 12 months after
  Proportion of participants that used the emergency department (ED) or had a treat and release ED or observation room visit and number of visits by study arm
Proportion of hospital admissions | 2 years before study start until 12 months after
  Proportion of participants who were hospitalized at least once and count of total hospitalizations from baseline to 12 months by study arm
Proportion of hospital readmissions | 2 years before study start until 13 months after
  Proportion of participants who were re-hospitalized within 30-days of the index hospitalization by study arm
Number of outpatient visits | 2 years before study start until 12 months after
  Number of primary care provider, specialist, mental health, and addiction medicine visits across the 12 month study period by study arm
Change in self-rated physical and mental health | Baseline, 12 months
  Measured as the change in self-rated overall, physical, and mental health reported on a 0 to 5-response (excellent to poor) scale by study arm. Higher score corresponds to better self-rated health

OTHER OUTCOMES:
Change in proportion of participants with low food security | Baseline, 12 months
  Measured as the change in the proportion of participants with low food security. Low food security will be defined as one or more item answered with "Often true" in the Hunger Vital Sign. Change in proportion of participants with low food security, from baseline to 12 months
Change in why participants could not/did not eat healthy foods | Baseline, 12 months
  Measured using the 14-response options providing reasons why respondents have difficulty eating or not eating healthy foods
Change in self-reported number of health visits | Baseline, 12 months
  Measured based on the change in self-reported hospitalizations, doctors visits, and ED visits within the past 12 months measured as continuous outcome between 0 and 100 or more
Change in prevalence of social risks | Baseline, 12 months
  Measured using the change in severity or presence of other social risks assessed using validated survey items for housing insecurity, transportation barriers, and financial strain
Change in frequency and severity of trade-offs | Baseline, 12 months
  Measured using the proportion of participants who report sometimes or often making trade offs between paying for food and paying for medications or medical care, utilities, rent or mortgage, transportation, and education
Change in Patient-Reported Outcomes Measurement Information System 10-item (PROMIS-10) physical and mental health scale | Baseline, 12 months
  Measured using the validated 10-item measure (PROMIS-10) to assess self-rated health, quality of life, mental and physical health, social satisfaction, ability to carry out roles, ability to carry out everyday physical activities, experiences of fatigue, frequency of emotional problems, and average pain. Analysis will assess change in overall measure by study arm
Change in cost-based primary care use | Baseline, 12 months
  Measured using a 5-response question (never to often) to delays to medical care because of cost where often is a worse outcome.
Change in perceived stress | Baseline, 12 months
  Measured using changes in self-report based on a validated, 4-item perceived stress scale (PSS-4); scores range from 0-16 and higher scores correspond to higher perceived stress
Change in general self-efficacy | Baseline, 12 months
  Measured using changes in participant responses across the 10-item validated self-efficacy scale; scores range from 10-40 with higher scores corresponding to higher perceived general self-efficacy
Change in chronic disease self-efficacy | Baseline, 12 months
  Measured using changes in participant responses across the validated, two-item chronic disease self-efficacy scale; scores range from 1 to 10 with higher scores relating to higher chronic disease self-efficacy
Change in utilization characteristics | 2 years before study start until 12 months after.
  Measured using claims data to analyze utilization characteristics e.g., length of stay (total days, average number of days per stay), and days until next admit across the 12-month study period
Change in self-reported medication adherence | Baseline, 12 months
  Measured as an affirmative response to cost-based medication nonadherence; change measured as a negative to affirmative or vice-versa response from baseline by study arm
Change in claims-based medication adherence | 2 years before study start until 12 months after
  Measured using medical claims data and calculated based on daily supply
Change in claims-based medication count | 2 years before study start until 12 months after
  Measured in the medical claims as the total number of medications that the participant had at baseline and across the 12-month study period
Change in HbA1c | Baseline, 12 months
  Change in self-reported HbA1c from baseline by study arm
Change in utilization costs | 2 years before study start until 12 months after
  Total cost of utilization across study period for inpatient and outpatient utilization
Change in self-reported days of medication adherence | Baseline, 12 months
  The change in a single-item question asking patients how many days (out of 7) they missed taking one of their medications. Changes in the number of days reported from baseline by study arm. More days corresponds to higher medication nonadherence

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Gottlieb, MD, MPH, Principal Investigator — University of California, San Francisco; Caroline Fichtenberg, PhD, Principal Investigator — University of California, San Francisco; Danielle Hessler Jones, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- Social Interventions Research and Evaluation Network (SIREN), University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
These data are available to researchers at SIREN (UCSF) via a data use agreement and cannot be shared without authorization and release of information by the data's owners (Covered California).